CLINICAL TRIAL: NCT01890395
Title: Bioenergetics in Surgical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, William Richards, Principal investigator, University of South Alabama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-294
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Mitochondrial DAMP Levels in Surgical Patients
Keywords: mitochondrial DAMPS
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood collection (Other): procedure: Blood draws as the intervention
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — Blood sampling collected at 9 timepoints: pre-operative, during surgery X 3, immediately after surgery, 24 hrs post-op, 72 hrs post-op, 5 days and 7 days post

SUMMARY:
To identify patients who may be predisposed for developing MOF (multiple organ failure)by the sampling of blood.

DETAILED DESCRIPTION:
The rationale for doing this study is the recognition that mitochondrial DNA Damage Associated Molecular Patterns (mtDAMPs) accumulate in the circulation after severe injury. Furthermore our own studies in severely injured patients identify that the mtDAMPS are increased 3-28 fold in those patients who eventually develop multiple organ dysfunction syndrome (MODS) compared to those severely traumatized patients who did not develop MODS. The relative risk of death from MODS after severe trauma was increased 8-20 times in those patients with elevated mt DAMP levels.

This study is then being done to correlate mitochondrial damp levels in surgical trauma to assess the time course and the levels of mtDAMPs with the type of surgical procedure. We believe that this information will help us to determine the time course of events and the triggers for development of multiple organ dysfunction seen after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients @ USAMC undergoing surgical operations expected to have microcirculatory changes, i.e., CABG, open heart, aortic or other revascularizing operations, general surgical operations such as colon resections, bowel resections or any other surgical procedures in which the subject could be expected to or might develop multiple system organ failure.

Exclusion Criteria:

N/A

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
correlation mitochondrial damps (mDAMPS) and multiple organ system failure | 1 year
  Preliminary studies (at University of South Alabama)in the trauma and burn patients indicate that the level of mitochondrial damps are highly correlated with non-survival; that is, they reflect a massive trauma. They also reflect patients that have a propensity to go into multiple system organ failure. We believe that these measurements in our surgical patients will also reveal many of the same correlations with the correlation between microvascular circulation and the mitochondrial damps.

CONTACTS AND LOCATIONS:
Overall Officials: William O. Richards, MD, Principal Investigator — University of South Alabama, Department of Surgery
Locations (1):
- University of South Alabama Medical Center, Mobile, Alabama, United States